CLINICAL TRIAL: NCT04666142
Title: The Effect of Light on Sleep Quality and Physiological Parameters in Individuals in Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Kübra Pamuk, Principal Investigator- nurse, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: U1111-1260-6250; Kübra pamuk (Other: Istanbul University-Cerrahpasa)
Record Dates: First submitted 2020-11-11; First posted 2020-12-14 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-11

CONDITIONS: Sleep; Light
Keywords: Sleep Quality; Light; Intensive Care Unit
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: According to the results of randomization, the group to which the lighting system will be applied was assigned as "experiment", and the group that will continue standard ICU lighting as "control"
Who Masked: Participant
Masking Description: The principle of "loyalty and confidentiality" was adhered to by assuring individuals that their identities and personal information obtained from them would not be disclosed to anyone other than the researcher or that the information would not be allowed to be accessed by anyone other than the intended purpose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Individual Characteristics of the Individuals in the Experimental and Control Groups (Active Comparator): The personal characteristics of the individuals included in the study were examined.
  Interventions: Other: Comparison of the personal characteristics of the experimental and control groups
- Disease Characteristics of the Individuals in Experimental and Control Groups (Active Comparator): The intensive care experience of the individuals included in the study, their status of receiving respiratory support, and the reason for staying in the intensive care unit were explained.
  Interventions: Other: Comparison of the personal characteristics of the experimental and control groups
- Distribution of Findings Regarding Sleep Activity of the Individuals in Both Groups (Active Comparator): The personal characteristics of the individuals in the experimental and control groups regarding sleep were examined.
  Interventions: Other: Comparison of the personal characteristics of the experimental and control groups
- Comparison of the Individuals in the experimental and control groups after 24 hours of sleep (Active Comparator): The effect of light after 24 hours in the experimental and control groups of individuals hospitalized in the intensive care unit was examined.
  Interventions: Other: Light applied experimental group, control group treated with standard intensive care lighting
- Comparison of physiological parameters of individuals in both groups after 24 hours (Active Comparator): Comparison of the physiological parameters of the individuals in the experimental and control groups 24 hours after their admission to the ICU.
  Interventions: Other: Light applied experimental group, control group treated with standard intensive care lighting
- Comparison of the Sleep Times of the Individuals in Both Groups 48 Hours After Intensive Care (Active Comparator): The effect of light after 48 hours in the experimental and control groups of individuals hospitalized in the intensive care unit was examined.
  Interventions: Other: Light applied experimental group, control group treated with standard intensive care lighting
- Comparison of physiological parameters of individuals in both groups after 48 hours (Active Comparator): Comparison of the physiological parameters of the individuals in the experimental and control groups 48 hours after their admission to the ICU.
  Interventions: Other: Light applied experimental group, control group treated with standard intensive care lighting
- Distribution of Total Sleep Times of the Individuals in the Experimental and Control Groups (Active Comparator): The sleep times of the individuals in both groups were compared
  Interventions: Other: Light applied experimental group, control group treated with standard intensive care lighting

INTERVENTIONS:
Other: Comparison of the personal characteristics of the experimental and control groups — General characteristics of the individuals in the experimental and control groups were compared.
  Arms: Disease Characteristics of the Individuals in Experimental and Control Groups; Distribution of Findings Regarding Sleep Activity of the Individuals in Both Groups; Individual Characteristics of the Individuals in the Experimental and Control Groups
Other: Light applied experimental group, control group treated with standard intensive care lighting — According to the results of randomization, the group to which the lighting system will be applied was assigned as "experiment", and the group that will continue standard ICU lighting as "control"
  Arms: Comparison of physiological parameters of individuals in both groups after 24 hours; Comparison of physiological parameters of individuals in both groups after 48 hours; Comparison of the Individuals in the experimental and control groups after 24 hours of sleep; Comparison of the Sleep Times of the Individuals in Both Groups 48 Hours After Intensive Care; Distribution of Total Sleep Times of the Individuals in the Experimental and Control Groups

SUMMARY:
The research was carried out in randomized controlled experimental type in order to determine the effect of light in ICU on patients' sleep quality and physiological parameters. The cases were assigned to the experimental and control groups according to the simple randomization method.

The research universe; Between May 2019 and December 2019, sick individuals who were admitted to the 5 isolation rooms in the Reanimation Intensive Care clinic in the education and research hospital in Istanbul were formed. The research sample is; As a result of the power made for the study to be experimentally designed; a total of 148, with a minimum of 74 for each group. In collecting data; Patient Information Form, Numerical Pain Rating Scale, Richards Campbell Sleep Scale, Glaskow Coma Scale, Richmond Agitation Sedation Scale, Bedside Monitors were used to measure physiological parameters. The data obtained as a result of the research were made using the package program named SPSS (IBM SPSS Statistics 24).

DETAILED DESCRIPTION:
Sleep causes temporary, partial and periodic interruption of the organism's interaction with the environment, is a physiological condition that affects many systems. That sleep activity is a vital and important activity for individuals.They emphasized and sleep; the alternating state of inertia and inertia, around the human a situation where they do not respond to the events that took place. initiation and maintenance through the function of many cortical and subcortical brain regions. People sleep on average one third of their lives They spend it. The sleep of a normal adult person consists of night sleep and It lasts an average of 7 to 9 hours, with a sleep time of four to six 90 to 100 minutes. Non-REM (NREM) and REM sleep change cyclically. In the sleep-wake cycle in man, the most basic and determinant is the circadian rhythm. Circadian The rhythm refers to changes in the physiological and biological processes of the organism for about a day. The main center that regulates the circadian rhythm is located in the anterior hypothalamus as a double structure. suprachiasmatic nucleus (SKN). Light is the most important rhythm editor. Other regulators are social and are physical activities. Florence Nightingale and Virgina Henderson in love and day rhythm; defined the patient as two important factors in supporting the health of the individual. In the regulation of the circadian rhythm, the light and dark cycle in the external environment is important. The synthesis and release of melatonin is stimulated in the dark at night, and during the day by the effect of light It is suppressed. N-acetyl transferase (NAT) enzyme is effective in melatonin formation. Melatonin The main task of the hormone is to protect the biological rhythm of the body. In this context; lighting, circadian rhythm and sleep are related.

Health care institutions and especially intensive care units, in terms of physical environment and lighting the patient can affect the circadian rhythm of the individual, change the release of melatonin and as a result can affect sleep patterns and cognitive performance. In our country, in terms of physical environment lighting, it does not support circadian rhythms. As a result, sick individuals in the ICU are asleep The therapeutic effect of sleep because they spend a significant amount of time they need to be awake can not benefit sufficiently. In addition, in the ICU, many There is a factor. These factors are; pain, physical condition, drug therapy, fear of death, environmental noise, pleasant non-smells, invasive interventions, loss of privacy and family disability. In the study of, the greatest stress of the sick individuals in the ICU One of the causes was found to be sleeping problems. In the literature, especially in health care institutions In patients with ICU inpatient, sleep activity has a negative effect on both duration and quality. shows that it is affected In admission to the ICU, when environmental factors are not suitable, the patient especially the sleep activity of the individual is impaired and this process occurs even after the patient is discharged from YBU, can continue. One of the biggest reasons for this; Physical environment and lighting of ICUs in terms of disruption of circadian rhythms of sick individuals. The presence of night light suppresses the level of melatonin, which is normally the highest at night. Melatonin level is accepted as an indicator of circadian rhythm. Artificial lighting is a known factor in the disruption of the circadian rhythm. Sick individuals in the ICU, 24 hours it is exposed to artificial light throughout a cycle. Artificial lighting, health of the sick individual health care to help professionals continue their care and treatment practices It is applied at high levels for 24 hours in institutions such as ICU. Its as a result, daylight is often obscured / eliminated in ICUs and artificial lighting are added. Researches conducted, unnatural night disruption of circadian rhythms with illumination causes health problems related to sleep activity. It is also sufficient and relaxing non-sleep, negatively affects the immune system, wound healing process and cognitive functions of the sick individual. It affects in the same direction, increases the level of stress and delays its recovery. Sick individuals in the ICU are concerned with serious illnesses or injuries and care and treatment. The illness of the symptoms lies. Today, long-term health of an illness or injury in an ICU It is known to cause problems. Some of these problems are sleep problems due to lighting and circadian rhythm disturbances. our Country Study to determine the effect of environmental factors related to lighting on sleep problems in ICU There is. Nurses who continue the care and treatment of sick individuals in ICU, diagnosing problems early, identifying primary nursing diagnoses, existing stressors important role such as reduction, ensuring the necessary environmental regulation to create a therapeutic environment, and they have responsibilities. In this context, this research is based on YBU. to determine the effect of light on sleep quality and physiological parameters in individuals and nursing will be carried out to guide its applications.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* Not having a problem in terms of consciousness and sense organs
* A score of 9 or above on the Glaskow Coma Scale (GCS),
* Richmond Agitation-Sedation Scale (RASS) score was determined as -1,0,1.

Exclusion Criteria:

* Be under the age of 18
* Having a problem in terms of consciousness and sense organs,
* A GCS score below 9,
* Receiving inotropic support,
* Being fully sedated,
* Having a chronic disease such as chronic heart disease, dementia, psychosis,
* Identified as having severe brain injury.

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-12-28 (Actual)

PRIMARY OUTCOMES:
Change in sleep time with light intervention in experimental and control groups in the intensive care unit | After the patient was admitted to the intensive care unit, 48 hours of sleep time was recorded.
  A recirculating lighting system was installed in the isolation room for the experimental group in line with evidence-based design principles. Light fixture 120 cm from the floor. high and light shining up. The system was set up to operate at varying levels of 9 lights, illumination for 24 hours. No application other than the standard lighting system of the ICU was applied to the individuals in the control group. Actiwatch device was placed on the arm of the sick individuals. Thanks to this device, the sleep time of the individuals was recorded.

SECONDARY OUTCOMES:
The effect of light on the patient's systolic and diastolic blood pressure in the experimental and control groups in the intensive care unit. | The systolic and diastolic blood pressure of the patient who was admitted to the intensive care unit was recorded for 48 hours.
  The systolic and diastolic blood pressure of the individual was recorded hourly by the investigator through the bedside monitoring system for 48 hours after admission to the ICU.
The effect of light on patient's heart rate in intensive care unit in experimental and control groups. | The heart rate of the patient, who was admitted to the intensive care unit, was recorded for 48 hours.
  The heart rate of the individual was recorded hourly by the researcher through the bedside monitoring system for 48 hours after admission to the ICU.
The effect of light on patient's respiratory rate in intensive care unit in experimental and control groups. | The respiration of the patient who was admitted to intensive care unit was recorded for 48 hours.
  The respiration of the patient was recorded hourly by the researcher through the bedside monitoring system for 48 hours after admission to the ICU.
The effect of light on the patient's body temperature in the intensive care unit in the experimental and control groups. | The body temperature of the patient who was admitted to intensive care unit was recorded for 48 hours.
  The body temperature of the patient was recorded hourly by the researcher through the bedside monitoring system for 48 hours after admission to the ICU.

CONTACTS AND LOCATIONS:
Overall Officials: kübra pamuk, graduate, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul Education Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No